CLINICAL TRIAL: NCT06001593
Title: Pilot Study of Modulating Auditory Symptoms and Vertigo of Meniere's Disease by Non-invasive Mastoid Electric Stimulation: Double-blind, Randomized, Sham-controlled, Investigator-initiated Trial
Brief Title: Modulating Auditory Symptoms and Vertigo of Meniere's Disease by Non-invasive Mastoid Electric Stimulation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2304-098-1425
Record Dates: First submitted 2023-07-24; First posted 2023-08-21 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-07

CONDITIONS: Meniere's Disease
Keywords: Electrical stimulation; Electroceutical; Meniere's disease
MeSH Terms: conditions — Meniere Disease | interventions — Betahistine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- electircal stimulation + betahistine (Experimental)
  Interventions: Device: YPS-201b; Drug: betahistine
- sham electircal stimulation + betahistine (Sham Comparator)
  Interventions: Drug: betahistine; Device: YPS-201b
- betahistine (Other): control group
  Interventions: Drug: betahistine

INTERVENTIONS:
Device: YPS-201b — electrical stimulation device.
  Arms: electircal stimulation + betahistine
Drug: betahistine — Relieve symptoms of balance disorders or dizziness
Device: YPS-201b — sham electrical stimulation device.
  Arms: sham electircal stimulation + betahistine

SUMMARY:
This study is a Double-blind, Randomized, Sham-controlled, Investigator-initiated trial. To explore the effectiveness of non-invasive inner ear electrical stimulation of the mastoid behind the ear in controlling auditory symptoms and dizziness in patients with Meniere's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dizziness (Meniere's) only, who understand the nature of the study and are willing to participate voluntarily.
* The frequency of the hearing loss is between 250 kHz and 1 kHz.
* Patients with bilateral 500, 1000, and 2000 Hz hearing threshold averages within 65 dB HL
* Patients who have received conventional pharmacotherapy for other dizziness conditions with a washout period of 2 months.
* To be eligible for subjects in the active phase of the disease, there must be at least 1 vertigo attack in the 6 months before study entry.
* If tests for renal function, electrolytes, etc. are performed and no problems are found

Exclusion Criteria:

* Patients with an otologic condition other than Meniere'ss (dizziness) (otitis media, profound hearing loss, hyperacusis, etc.).
* Patients' conditions that may affect EEG measurements, such as a stroke, brain hemorrhage, or brain tumor.
* Patients with kidney disease
* Patients Have or have had a serious medical condition, such as cancer (including leukemia, blood cancers, epilepsy, and neuropsychiatric conditions).
* Patients with an artificial implant in the body (cochlear implant, hip joint, pacemaker, etc.)
* Women of childbearing potential, pregnant women, or nursing mothers
* Patients who can have Injuries or dermatologic abnormalities at the site of application of the equipment.
* Patients with coronary artery disease, uncontrolled high blood pressure, or other serious medical conditions (including kidney disease).

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Valuation of dizziness with Dizziness Visual Analogue scale(Efficacy) | 0,2,4,8,12 weeks during electrical stimulation
  Verifying therapeutic effect of electrical stimulation
Evaluate vestibular-ocular reflex with Video head impulse test(Efficacy) | 0,4,8,12 weeks during electrical stimulation
  Verifying therapeutic effect of electrical stimulation,evaluate the function of the vestibulocochlear reflex in the semicircular canal and measure the extent of improvement in Meniere's disease.
Valuation of hearing threshold with pure tone audiometry(Efficacy) | 0,4,8,12 weeks during electrical stimulation
  Verifying therapeutic effect of electrical stimulation.measuring the level of enhancement in low-frequency hearing.
electroencephalography(Efficacy) | 0,1,4,8,12 weeks during electrical stimulation
  Verifying therapeutic effect of electrical stimulation,evaluate the inhibitory response of the brain through EEG readings following repeated stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No